CLINICAL TRIAL: NCT01885819
Title: Feasibility Study of Non-Expanded Autologous Adipose Tissue Derived Stromal Vascular Fraction Cells in Disease Modifying Anti-Rheumatic Drugs (DMARD) Resistant Rheumatoid Arthritis
Brief Title: Autologous Adipose Tissue Stromal Vascular Fraction Cells for Rheumatoid Arthritis
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: per sponsor decision
Sponsor: Translational Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TBS-SVF-AR-002-2013
Record Dates: First submitted 2013-06-18; First posted 2013-06-25 (Estimated); Last update posted 2017-08-10 (Actual); Status verified 2017-08

CONDITIONS: Rheumatoid Arthritis
Keywords: Adipose stromal vascular fraction; Rheumatoid arthritis; adult stem cells
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (Experimental): Autologous stromal vascular fraction cells
  Interventions: Biological: Autologous stromal vascular fraction cells

INTERVENTIONS:
Biological: Autologous stromal vascular fraction cells

SUMMARY:
Autologous stromal vascular fraction (SVF) injected at 8 and 10 days after extraction is safe and useful procedure in inducing remission of RA in patients resistant to standard DMARD therapy.

DETAILED DESCRIPTION:
The proposed study will assess primarily safety and secondary efficacy endpoints of autologous stromal vascular fraction (SVF) cells administered to 20 patients with disease modifying antirheumatic drug (DMARD)-resistant Rheumatoid Arthritis (RA) who have been nonresponsive to at least one course of one DMARD selected from a group comprising of: gold salts, leflunomide, methotrexate, and hydroxychloroquine.

The primary objective of safety will be defined as freedom from treatment associated adverse events for the period of one year. The secondary objective of efficacy will include evaluation at baseline and at months 1, 2, 3 and 6 of efficacy endpoints of CRP, ESR, anti-citrulline antibody, RF, Quality of Life Questionnaire, 28-joint disease activity score (DAS28), European League against Rheumatism (EULAR) response criteria and immunological parameters.

ELIGIBILITY:
Inclusion Criteria:

Age older than 18 years and ability to understand the planned treatment.

Patients of either gender with RA with a duration of 6 to 72 months defined as the presence of at least three of the following criteria: 6 or more painful, 2 or more swollen joints, morning stiffness for at least 45 minutes (on average during the week prior to entry), and an erythrocyte sedimentation rate (ESR) of at least 28 mm.

Nonresponsive to at least one course of one DMARD selected from the group comprising of: gold salts, leflunomide, methotrexate, and hydroxychloroquine.

Second-line agents are discontinued at least 4 weeks prior to entry.

Able to tolerate ALL study procedures

Able to give informed Consent

Negative for HcG with a serum pregnancy test

Hematocrit ≥ 28.0%, White Blood Cell count ≤ 14,000, Platelet count ≥ 50,000,

Life expectancy of 6 months or more in the opinion of the investigator

Serum bilirubin, ALT, AST up to 2.5 time the upper level of normal.

Controlled blood pressure (systolic blood pressure ≤140 and a diastolic blood pressure of ≤90 mmHG) and established anti-hypertensive therapy as necessary prior to entry into the study

Patient has received stable, standard medical therapy for at least one month with no new medications to treat the disease introduced in the last month.

Pre-existing condition (e.g. thromboembolic risk, diabetes, hypercholesterolemia) are adequately controlled in the opinion of the investigator

Fertile patients (male and female) must agree to use an appropriate form of contraception while participating in the study.

Exclusion Criteria:

Female who is pregnant or nursing, or of child bearing potential and is not using a reliable birth control method, or who intend to become pregnant during the tenure of this study.

History of prior radiation exposure for oncological treatment.

History of Bone Marrow Disorder (especially NHL, MDS)

History of abnormal bleeding or clotting.

History of Liver Cirrhosis.

End stage renal disease (Creatinine ≤ 3.0 mg / dl) and/or dialysis

Active clinical infection being treated by antibiotics before one week enrollment

Inability or unwillingness to comply with the treatment protocol, follow-up, research tests, or give consent.

History of life-threatening arrhythmias, except if an automated implantable cardioverter defibrillator (AICD) is implanted

Life expectancy <6 months due to concomitant illnesses

Known cancer and undergoing treatment; chemotherapy and/or radiotherapy

Patients receiving treatment with hematopoietic growth factors (e.g., EPO, G-CSF)

Patients who can not stop anticoagulation therapy (warfarin) 72hrs prior to infusion

Patients who can not stop anti-platelet therapy (clopidogrel) 7 days prior infusion Prior admission for substance abuse

Body Mass Index (BMI) of 40 kg/m2 or greater

Patient receiving experimental medication or participating in another clinical study within 30 days of signing the informed consent

In the opinion of the investigator or the sponsor, the patient is unsuitable for cellular therapy

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-06; Primary Completion 2016-07 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events | 6 months

SECONDARY OUTCOMES:
Change from baseline 28-DAS Score at 6 months | 6 months
Change from baseline EULAR Response Criteria at 6 months | 6 months
  Change in European League against Rheumatism (EULAR) response criteria and immunological parameters from baseline to 6 months.
Change from baseline quality of life measure (based on Stanford HAQ) at 6 months | 6 months
Change from baseline C-reactive protein at 6 months | 6 months
Change from baseline erythrocyte sedimentation rate (ESR) at 6 months | 6 months
Change from baseline anti-citrulline antibody measure at 6 months | 6 months
Change from baseline rheumatoid factor (RF) at 6 months | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Paz-Rodriguez, MD, Principal Investigator — Stem Cell Institute
Locations (1):
- Stem Cell Institute, Panama City, Panama